CLINICAL TRIAL: NCT06720246
Title: Effects of Bariatric Surgery and Pharmacological Therapy with Liraglutide on Motivational and Inhibitory Processes: Cognitive-Behavioral Markers of Long-Term Weight Loss. a Study on Patients with Obesity.
Brief Title: Impact of Bariatric Surgery and Liraglutide on Cognitive-Behavioral Markers of Long-Term Weight Loss in Obesity
Acronym: Balance
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: BALANCE; RC2024 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Overweight
Keywords: Obesity; Bariatric surgery; food cognition; liraglutide
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bariatric Surgery: Patients submitted to bariatric surgery
- Liraglutide: Patients submitted to liraglutide treatment

SUMMARY:
The present research project aims to study the effects of bariatric surgery and liraglutide administration (in patients already selected for one of these procedures) on two cognitive-behavioral processes partially supported by distinct brain networks: automatic approach tendencies (underpinned by the cue-reactivity network) and behavioral inhibition (underpinned by the cue-regulation network). Additionally, the investigators aim to study how these processes may be modulated by satiety. The secondary objective of the project includes identifying cognitive-behavioral markers that can predict the response to these treatments.

DETAILED DESCRIPTION:
Experimental and meta-analytic neuroimaging studies have highlighted two primary brain networks whose functioning or structure is altered in patients with obesity: (i) the "cue-reactivity network," involved in sensory, hedonic, and motivational responses to food, and (ii) the "cue-regulation network," more prominently involved in attentional, decision-making, and inhibitory processes. In line with this theoretical framework, weight loss induced by pharmacological treatments or bariatric surgery is associated with a partial recovery of the functioning and structure of these brain networks.

Following a sleeve gastrectomy, obese patients exhibit reduced activity in the reward circuit and increased activity in the inhibitory control circuit in response to high-calorie food images, suggesting a normalization of brain responses to food after bariatric surgery. Moreover, these changes in brain functionality may be accompanied by increased gray matter density in the prefrontal cortex, which persists for up to 12 months following sleeve gastrectomy or Roux-en-Y gastric bypass.

Pharmacologically, the administration of glucagon-like peptide-1 receptor (GLP-1) agonists-such as liraglutide, semaglutide, and exenatide-has proven effective in treating diabetes and promoting weight loss. fMRI studies have shown that intravenous administration of exenatide (vs. placebo) in patients with obesity and type 2 diabetes reduces neurofunctional activity in key nodes of the cue-reactivity network (e.g., amygdala, putamen, insula) in response to high-calorie food images. Furthermore, this effect is nullified if exenatide administration is preceded by GLP-1 receptor blockade.

However, it remains unclear whether such surgical or pharmacological treatments are accompanied by changes in cognitive processes associated with reactivity to edible stimuli or behavioral inhibition, and whether these contribute to an improved post-operative response to satiety.

This research project thus aims to study the effects of bariatric surgery and liraglutide administration (in patients already selected for one of these procedures) on two cognitive-behavioral processes partially supported by distinct brain networks: automatic approach tendencies (underpinned by the cue-reactivity network) and behavioral inhibition (underpinned by the cue-regulation network). Additionally, the investigators aim to study how these processes may be modulated by satiety. The secondary objective of the project involves identifying cognitive-behavioral markers that could predict responses to these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any ethnicity, aged between 20 and 60 years.
* BMI equal to or greater than 30 kg/m².
* No history of neurological or psychiatric disorders, as confirmed through medical history and neuropsychological screening.
* Signed informed consent and willingness to comply with all study procedures.
* Patients scheduled for surgery, treatment with liraglutide, or a dietary regimen.

Exclusion Criteria:

* Previous diagnosis of significant neurological conditions (e.g., brain injury or dementia) or major psychiatric disorders.
* Current or past psychopharmacological therapy, if prolonged.
* BMI lower than 30 kg/m².
* Lack of signed informed consent.
* Severe medical conditions, including but not limited to: hypertension, significant cardiac disease, or other disorders that may compromise patient safety.
* Confirmed pregnancy through self-report and/or breastfeeding.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited at the IRCCS Galeazzi-Sant'Ambrogio, Milan.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Reaction times (approach bias) | Baseline and after treatment (2-4 months)
  Changes in reaction times (approach bias) in response to pictures of high-calorie and low-calorie foods after treatment.
Accuracy (inhibition) | Baseline and after treatment (2-4 months)
  Changes in accuracy (inhibition) in response to high-calorie and low-calorie food pictures after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No